CLINICAL TRIAL: NCT03218605
Title: Effect of Warming-up Activities on the Vascularisation of the Achilles Tendon: a Cohort Study
Brief Title: Which Physical Activity Influences Achilles Tendon Blood Flow the Most?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013/401
Record Dates: First submitted 2017-07-05; First posted 2017-07-14 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Physical Activity
Keywords: Achilles tendon; Warming-up; Vascularisation; Physical activity; Oxygen-to-See (O2C)
MeSH Terms: conditions — Motor Activity; Neovascularization, Pathologic | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy active participants (Experimental)
  Interventions: Other: physical activity

INTERVENTIONS:
Other: physical activity — Subjects performed five activities: running, static stretch, dynamic stretch, cycling and rope skipping

SUMMARY:
Previous studies have shown that a decreased blood flow is a risk factor in the occurrence of Achilles tendon (AT) injuries. Based on the current literature, no consensus was reached as to the most solid warming-up of the AT. Therefore, knowledge about activities which increase blood flow in the AT could be useful in the development of a solid warming-up programme for the AT. The aim of this investigation was to define the influence of different kinds of physical activity on the vascularisation of the AT in a healthy asymptomatic population. Subjects performed five activities in randomized order: running, static stretch, dynamic stretch, cycling and rope skipping. The vascularisation of the AT of the dominant limb was measured with the non-invasive oxygen-to-see (O2C) device. Blood flow was measured before, immediately after, five and ten minutes after activity to investigate the duration of the vascular response to activity.

ELIGIBILITY:
Inclusion Criteria:

* no history of Achilles tendon complaints
* healthy and active adolescents

Exclusion Criteria:

* history of Achilles tendon pain or current complaints
* not healthy or not active population
* children

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Achilles tendon blood flow | 3 minutes before and immediately (0 minutes) after the physical activity to assess the change in blood flow due to the physical activity
  measured with the non-invasive O2C device

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wezenbeek E, De Clercq D, Mahieu N, Willems T, Witvrouw E. Activity-Induced Increase in Achilles Tendon Blood Flow Is Age and Sex Dependent. Am J Sports Med. 2018 Sep;46(11):2678-2686. doi: 10.1177/0363546518786259. Epub 2018 Aug 1. PMID 30067065